CLINICAL TRIAL: NCT06374199
Title: A Pilot Study of a Food is Medicine Intervention to Improve Pregnancy Outcomes
Brief Title: Med-South Lifestyle Program for Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-0181
Record Dates: First submitted 2024-04-15; First posted 2024-04-18 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Pregnancy Complications
MeSH Terms: conditions — Pregnancy Complications

STUDY DESIGN:
Intervention Model Description: Standard 2 group parallel randomized trial study design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nuts and Extra Virgin Olive Oil (Active Comparator): Intervention includes lifestyle counseling and food provisions including extra virgin olive oil (EVOO) and nuts
  Interventions: Behavioral: Med-South Lifestyle Intervention for Pregnancy--Arm 1
- Nuts, Extra Virgin Olive Oil, and Medically Tailored Meals (Experimental): Intervention includes lifestyle counseling and food provisions including extra virgin olive oil (EVOO), nuts, and medically tailored meals
  Interventions: Behavioral: Med-South Lifestyle Intervention for Pregnancy--Arm 2

INTERVENTIONS:
Behavioral: Med-South Lifestyle Intervention for Pregnancy--Arm 1 — Intervention includes lifestyle counseling and food provisions including extra virgin olive oil and nuts
  Arms: Nuts and Extra Virgin Olive Oil
Behavioral: Med-South Lifestyle Intervention for Pregnancy--Arm 2 — Intervention includes lifestyle counseling and food provisions including extra virgin olive oil, nuts, and medically tailored meals
  Arms: Nuts, Extra Virgin Olive Oil, and Medically Tailored Meals

SUMMARY:
Eating a Mediterranean-style diet during pregnancy improves pregnancy outcomes, yet most Americans who are pregnant do not follow this type of dietary pattern. There is increasing interest in Food is Medicine programs, which provides foods to patients to improve health outcomes - food provided in this context is called medically tailored meals. The research team at the UNC Center for Health Promotion and Disease Prevention is developing a Food is Medicine program to improve pregnancy outcomes and at this point the team is ready to test the program.

The purpose of this study is to assess the feasibility and acceptability of a Food is Medicine intervention when started during the first trimester of pregnancy. The eating pattern to be evaluated in this study is a Mediterranean-style dietary pattern adapted for the southern United States - thus, the program is called "Med-South." All who take part will receive Med-South dietary counseling. In addition, to help participants follow a Med-style dietary pattern, one group of study participants will receive extra virgin olive oil and nuts. The other group will receive extra virgin olive oil, nuts, and frozen meals (medically tailored meals) that align with the Med-South dietary pattern. Participants will be assigned at random (like flipping a coin) to one of these groups

DETAILED DESCRIPTION:
For those taking part in this study, participation study will last from the enrollment visit (staring as early as possible during the 1st trimester, but < 15 weeks of pregnancy) to delivery-for most this will be about 24 weeks, but less for those who deliver early. There will be 10 counseling sessions throughout the study. Three sessions will be in-person and will include study measures. The other 7 sessions can be done over the phone or in person. Also, there are 4 optional phone counseling sessions. Each session will last approximately 10-45 minutes (except the first session, which may last an hour).

The risk of taking part in this study is minimal as the dietary pattern being tested is NOT experimental. This study is promoting a diet pattern that aligns with the United States Department of Agriculture (USDA) 2020-25 guidelines for people who are pregnant. A risk of all research studies is loss of confidentiality, but the study team will take all standard measures to reduce this risk.

In terms of benefits, if one takes part in this study and follows the dietary recommendations, pregnancy outcomes may be improved. Also, the food received as part of this study may be considered a benefit.

Both intervention groups will receive nuts and olive oil valued at $50 per month for up to 6 months (time of delivery). Participants in the group that only receives olive oil and nuts will also receive a grocery store gift card each month for up to 6 months (or time of delivery) while those in the group receiving medically tailored meals will receive 7 frozen meals a week for up to 6 months (or time of delivery).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Patient plans to receive prenatal care at UNC OB/GYN at Weaver Crossing
* Patient deemed to have viable singleton pregnancy and approved for participation by OB clinician
* Gestational age < 15 weeks
* Patient able to consume nuts, EVOO, or both

Exclusion Criteria:

* Patient is not fluent in English
* Patient does not have access to internet by web, tablet, or smart phone
* Type 1 diabetes
* Pregnant with twins or a greater number of fetuses

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — The study will enroll participants who are pregnant whatever their gender identity.
Enrollment: 35 (Actual)
Dates: Start 2024-05-10 (Actual); Primary Completion 2025-07-05 (Actual); Study Completion 2025-07-05 (Actual)

PRIMARY OUTCOMES:
Percent that would recommend this program to others who are pregnancy | Assessed at approximately 24 and 36 weeks of pregnancy
  Percent who report they strongly agree or agree (other options on scale -- neither, agree, strongly disagree) with the statement: "I would recommend this program to others who are pregnant."
Percent of participants who take part in the 10 study counseling sessions | from enrollment to delivery (approximately 40 weeks of pregnancy)
  Percentage of participants who attend at 8 of the 10 sessions

SECONDARY OUTCOMES:
Maternal diet quality | Assessed at approximately 24 and 36 weeks of pregnancy
  Quality of diet during pregnancy assessed with modified Prevención con Dieta Mediterránea (PREDIMED) study screener. The modified PREDIMED screener consists of 12 items, each scored as healthful or not (1 for healthful and 0 for not healthful), with items summed for a total score.

OTHER OUTCOMES:
skin carotenoids | Assessed at approximately 24 and 36 weeks of pregnancy
  Assessed by Reflection Spectroscopy Device ("Veggie Meter"™). Results is a score that reflects skin carotenoid content with is correlated with fruit and vegetable intake. The score is assessed 3 times and averaged.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Keyserling, MD, Principal Investigator — University of North Carollina at Chapel Hill
Locations (1):
- Center for Health Promotion and Disease Prevention/UNC-Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No